CLINICAL TRIAL: NCT04568954
Title: Molbio Truenat TB Platform Combined With the Truenat TB Assays for Detection of Tuberculosis and Rifampicin Resistance in Adults With Presumptive Pulmonary Tuberculosis at Primary-level Diagnostic Centres in Tanzania and Mozambique: a Pragmatic, Cluster-randomized Controlled Trial
Brief Title: TB-CAPT CORE Truenat Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); National Institute for Medical Research, Tanzania (Other Government); Centro de Investigação em Saúde de Manhiça (Other); Instituto Nacional de Saúde, Mozambique (Other Government); Ifakara Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TB041-3/1
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis; Diagnoses Disease
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The objective of the trial is to assess Truenat platform/TB assays in clinical care. The use of Truenat platform/TB assays does not allow blinding of clinicians and participants in this trial. The trial-related procedures will be embedded into the routine practice at the primary-level facility. Data analysts will be blinded to intervention allocation.
  Randomisation takes place on a cluster level rather than for the individual patients to avoid contamination between the arms within a health facility. Since clinics will be relatively far apart, contamination is unlikely.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TB testing using the Truenat platform/TB assays (Experimental): TB testing using the Truenat platform/TB assays placed at primary health care clinics combined with rapid communication of results and same day TB treatment initiation
  Interventions: Diagnostic Test: Truenat TB platform/TB assays
- Standard of care Arm (No Intervention): Standard of care for TB testing using a combination of smear microscopy and laboratory (off-site) Xpert testing, may vary by clinic depending on availability of transport and stock of Xpert MTB/RIF or Xpert MTB/RIF Ultra cartridges (Xpert).

INTERVENTIONS:
Diagnostic Test: Truenat TB platform/TB assays — Truenat TB platform/TB assays, a molecular diagnostic test developed by Molbio diagnostics, for the diagnosis of Mycobacterium tuberculosis complex (MTBC) and Truenat MTB-RIF Dx for detection of RIF resistance was endorsed in 2020 by the WHO for TB diagnosis.
  The system has been designed to be operated as a point-of-care- diagnostic solution in peripheral laboratories with minimal infrastructure.
  It takes about 25 minutes to do the DNA extraction and another 35 minutes to diagnose TB.
  It is portable and battery operated, have no need for a computer or laptop, and operate from 2-40 C ambient temperature. The system uses room temperature stable reagents with long shelf life.
  Arms: TB testing using the Truenat platform/TB assays

SUMMARY:
A cluster randomized controlled trial to evaluate the effect of placing Truenat platform/TB assays at primary health care clinics combined with rapid communication of results on time to treatment initiation of microbiologically confirmed TB.

DETAILED DESCRIPTION:
A cluster randomized controlled trial to evaluate the effect of placing Truenat platform/TB assays at primary health care clinics combined with rapid communication of results on time to treatment initiation of microbiologically confirmed TB.

In a setup period (survey of study centers) before randomization, the healthcare facilities (=clinics) of 4 sites will be asked to provide information about the number of TB notifications per quarter covering the period 1/2018-6/2020. From this information the foreseeable number of examined patients ("size of a clinic") will be derived, which will be used as a strata variable in randomization process.

Facilities will be randomly allocated to the standard of care (control), or Truenat platform/TB assays (intervention).

A cluster refers to a clinic. The clusters will be assigned to intervention or control arm to one of two diagnostic procedures (SOC [smear microscopy and/or Xpert MTB/RIF Ultra off-site] vs Truenat platform/TB assays on-site) following a restricted randomization strategy, whereby 6 to 8 strata of clusters will be established using the stratification variables site (clinics belong to a site) and size and apply balance criteria for them. The number of strata per site depends on heterogeneity of the sizes of the clinics as established in setup period and may be increased, typically 1 or 2 strata per site will be established.

The primary endpoint will be compared in an individual level analysis with strata and intervention as fixed effects and cluster as random effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients with presumptive pulmonary TB, as defined by the national TB treatment guidelines in each country: patients with cough more than 1-2 weeks and/or fever, night sweats, blood-stained sputum (haemoptysis) significant weight loss, abnormalities on chest radiograph
* Adults 18 years old and above who are able and willing to consent

Exclusion Criteria:

* Circumstances that raise doubt on free, informed consent (e.g. in a mentally impaired person or a prisoner)
* Already diagnosed with TB
* Currently receiving anti-TB therapy
* Patients with symptoms which are only attributable to extra-pulmonary TB
* Patients who are seriously ill and need to be admitted to hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3987 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with microbiological confirmation starting TB treatment within 7 days of their first visit among enrolled participants | 7 days
  Proportion of participants with microbiological confirmation starting TB treatment within 7 days of their first visit among enrolled participants

SECONDARY OUTCOMES:
Time to bacteriological confirmation of TB | 60 days
  Time to bacteriological confirmation of TB (up to 180 days) from enrolment
Proportion of patients treated for TB up to 60 days from enrolment | 60 days
  Proportion of patients treated for TB up to 60 days from enrolment
Proportion of participants with signs and symptoms suggestive of pulmonary TB starting TB treatment with microbiological confirmation within 60 days from enrolment | 60 days
  Proportion of participants with signs and symptoms suggestive of pulmonary TB starting TB treatment with microbiological confirmation within 60 days from enrolment
Cost and productivity related endpoints | 60 days
  Patients' costs related to care at 60 days from enrolment.
  * Number of lost working days over the past month at 60 days from enrolment
  * Monthly earning in the past month at 60 days from enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Kranzer, Principal Investigator — Medical Center of the University of Munich
Locations (4):
- Mozambique (2):
  - Centro de Investigação em Saúde de Manhiça-Fundação, Manhiça, Vila Da Manhiça
  - Instituto Nacional de Saúde (INS), Maputo
- Tanzania (2):
  - Ifakara Health Institute, Dar es Salaam
  - National Institute of Medical Research (NIMR), Mbeya

IPD SHARING:
Plan to Share IPD: Yes
Individual, de-identified participant data may be shared, including data dictionaries. Available documents include the study protocol and statistical analysis plan. Templates of the informed consent forms may be shared upon request. The data will be available immediately following publication with no end date, will be shared with anyone who wishes to access them, and will be available for any purpose of analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon publication of the main study manuscript

REFERENCES:
- [Derived] Inbaraj LR, Daniel J, Sathya Narayanan MK, Srinivasalu VA, Bhaskar A, Scandrett K, Rajendran P, Kirubakaran R, Shewade HD, Malaisamy M, Padmapriyadarsini C, Takwoingi Y. Truenat MTB assays for pulmonary tuberculosis and rifampicin resistance in adults and adolescents. Cochrane Database Syst Rev. 2025 Mar 24;3(3):CD015543. doi: 10.1002/14651858.CD015543.pub2. PMID 40122135
- [Derived] Leukes VN, Hella J, Sabi I, Cossa M, Khosa C, Erkosar B, Mangu C, Siyame E, Mtafya B, Lwilla A, Viegas S, Madeira C, Machiana A, Ribeiro J, Garcia-Basteiro AL, Riess F, Elisio D, Sasamalo M, Mhalu G, Denkinger CM, Castro MDM, Bashir S, Schumacher SG, Tagliani E, Malhotra A, Dowdy D, Schacht C, Buech J, Nguenha D, Ntinginya N, Ruhwald M, Penn-Nicholson A, Kranzer K; TB-CAPT Consortium. Study protocol: a pragmatic, cluster-randomized controlled trial to evaluate the effect of implementation of the Truenat platform/MTB assays at primary health care clinics in Mozambique and Tanzania (TB-CAPT CORE). BMC Infect Dis. 2024 Jan 19;24(1):107. doi: 10.1186/s12879-023-08876-8. PMID 38243223

DOCUMENTS (2):
  • Study Protocol (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT04568954/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT04568954/SAP_001.pdf